CLINICAL TRIAL: NCT00831012
Title: A Phase I Dose Comparison Study of the Safety and Immunogenicity of rDEN3delta30/31-7164, a Live Attenuated Virus Vaccine Candidate for the Prevention of Dengue Serotype 3
Brief Title: Safety of and Immune Response to a Dengue Virus Vaccine (rDEN3delta30/31-7164) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIR 257
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Dengue Fever
Keywords: Dengue Vaccine; Dengue Virus; Dengue Hemorrhagic Fever; Dengue Shock Syndrome
MeSH Terms: conditions — Dengue; Severe Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Group 1 will consist of healthy participants receiving an immunization of 10^3 PFU rDEN3delta30/31-7164
  Interventions: Biological: rDEN3delta30/31-7164
- Group 2 (Experimental): Group 2A will consist of healthy participants who will receive an immunization of 10^5 PFU of rDEN3delta30/31-7164 vaccine or placebo. Group 2A participants will be enrolled if less that 90% of Group 1 participants seroconvert to DEN3 by Study Day 42.
  Group 2B will consist of healthy participants who will receive an immunization of 10^1 PFU of rDEN3delta30/31-7164 vaccine or placebo. Group 2B participants will be enrolled if more that 90% of Group 1 participants seroconvert to DEN3 by Study Day 42.
  Interventions: Biological: rDEN3delta30/31-7164

INTERVENTIONS:
Biological: rDEN3delta30/31-7164 — A live attenuated, recombinant DEN3 candidate vaccine virus

SUMMARY:
Dengue fever, which is caused by dengue viruses, is a major health problem in tropical and subtropical regions of the world. The purpose of this study is to test the safety of and immune response to a new dengue virus vaccine in healthy adults.

DETAILED DESCRIPTION:
More than 2 billion people living in tropical and subtropical regions of the world are at risk of dengue virus infection. Dengue viruses cause dengue fever, as well as the more severe dengue hemorrhagic fever/shock syndrome, and dengue virus infection is the leading cause of hospitalization and death in children in several tropical Asian countries. This study will evaluate the safety and immunogenicity of a live, attenuated dengue virus called rDEN3delta30/31-7164.

This study will consist of two groups, with Group 1 enrolling first. Group 1 participants will be randomly assigned to receive either 10^3 PFU of rDEN3delta30/31-7164 or placebo subcutaneously in their deltoid. Participants will be monitored at the clinic for 30 minutes after receiving the immunization to monitor for adverse effects. After that, participants will be asked to return to the clinic approximately every other day for the next 16 days, and then on Day 21, 28, 42, and 180. At each visit participants will have physical and clinical exams, vital signs, measures, blood drawn, and will be asked about any adverse events they may have experience. Female participants will be given a pregnancy test. In addition, participants will be asked to measure their temperature 3 times a day and record it in a temperature diary for the first 16 days after immunization.

If less than 90% of the participants in Group 1 seroconvert to DEN3 then Group 2A will be enrolled. Group 2A will follow the same procedures as Group 1, but will receive a 10^5 PFU dose of rDEN3delta30/31-7164.

If more than 90% of the participants in Group 1 seroconvert to DEN3 then Group 2B will be enrolled. Group 2A will follow the same procedures as Group 1, but will receive a 10^1 PFU dose of rDEN3delta30/31-7164.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or non-pregnant female between 18 and 50 years of age, inclusive.
* Good general health as determined by physical exam, laboratory screening, and review of medical history
* Available for the duration of the study, approximately 26 weeks post-vaccination
* Willing to use effective means of contraception for the duration of the trial

Exclusion Criteria:

* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the volunteer to understand and cooperate with the requirements of the study protocol
* Grade 1 or above values for absolute neutrophil count (ANC), alanine aminotransferase (ALT), and serum creatinine, as protocol defined
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating n the trial or would render the volunteer unable to comply with the protocol
* Any significant alcohol or drug abuse in the past 12 months which has caused medical, occupational, or family problems, as indicated by volunteer history
* History of a severe allergic reaction or anaphylaxis
* Severe asthma (emergency room visit or hospitalization within the last 6 months)
* Positive HIV-1 serology by screening and confirmatory assays
* Positive for hepatitis C virus (HCV) by screening and confirmatory assays
* Positive for hepatitis B virus (HBV) by hepatitis B surface antigen (HBsAg) screening
* Any known immunodeficiency syndrome
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days prior to Study Day 0
* Receipt of a live vaccine within 4 weeks or a killed vaccine within the 2 weeks prior to Study Day 0 or anticipated receipt of any vaccine during the 42 days following Study Day 0
* History of a surgical splenectomy
* Receipt of blood products within the past 6 months, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 42 days following Study Day 0
* History or serologic evidence of previous dengue virus infection or other flavivirus infection (e.g., yellow fever virus, St. Louis encephalitis, West Nile virus)
* Previous receipt of yellow fever or dengue vaccine (licensed or experimental)
* Receipt of any investigational agent in the 30 days prior to Vaccination Day 0 or plan to participate in any investigational drug trials during the next 26 weeks
* Definite plans to travel to a dengue endemic area
* Pregnancy or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Determine the safety of a single dose of the rDEN3Δ30/31-7164 vaccine, as assessed by the frequency, severity, and seriousness of vaccine related adverse events (AEs). | Throughout study
Determine the immunogenicity of a single dose of the rDEN3delta30/31-7164 vaccine, as assessed by neutralizing antibody titers to DEN3 at 4 weeks and 6 weeks after vaccination | Throughout study

SECONDARY OUTCOMES:
Assess the frequency, quantity, and duration of viremia after a single dose of vaccine | Throughout study
Determine the number of vaccinees infected with rDEN3delta30/31-7164. Infection is defined as recovery of vaccine virus from the blood or serum of a volunteer and/or by seroconversion to DEN3 (a ≥4-fold rise in DEN3 neutralizing antibody titers). | Throughout study
Compare the infectivity rates, safety, and immunogenicity of a single dose of rDEN3delta30/31-7164 vaccine between the dose level groups. | Throughout study
Determine the durability of antibody response 26 weeks after vaccination | At 26 weeks
Obtain an estimate for the Human Infectious Dose-50% (HID50) if dose dependent infectivity is observed | Throughout study
Evaluate the phenotype of peripheral blood mononuclear cells at primary infection with the rDEN3delta30/31-7164 vaccine. | Throughout study
Evaluate the cellular and humoral immune response to primary infection with the rDEN3delta30/31-7164 vaccine | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Study Chair — Center for Immunization Research (CIR), Johns Hopkins School of Public Health
Locations (1):
- Center for Immunization Research, Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Popper SJ, Strouts FR, Lindow JC, Cheng HK, Montoya M, Balmaseda A, Durbin AP, Whitehead SS, Harris E, Kirkpatrick BD, Relman DA. Early Transcriptional Responses After Dengue Vaccination Mirror the Response to Natural Infection and Predict Neutralizing Antibody Titers. J Infect Dis. 2018 Nov 5;218(12):1911-1921. doi: 10.1093/infdis/jiy434. PMID 30010906
- [Derived] Katzelnick LC, Fonville JM, Gromowski GD, Bustos Arriaga J, Green A, James SL, Lau L, Montoya M, Wang C, VanBlargan LA, Russell CA, Thu HM, Pierson TC, Buchy P, Aaskov JG, Munoz-Jordan JL, Vasilakis N, Gibbons RV, Tesh RB, Osterhaus AD, Fouchier RA, Durbin A, Simmons CP, Holmes EC, Harris E, Whitehead SS, Smith DJ. Dengue viruses cluster antigenically but not as discrete serotypes. Science. 2015 Sep 18;349(6254):1338-43. doi: 10.1126/science.aac5017. PMID 26383952